CLINICAL TRIAL: NCT05967325
Title: Safety and Feasibility of Stromal Vascular Fraction (SVF) Combined With Functional Self-assembling Peptide Nanofiber Hydrogels in the Treatment of Spinal Cord Injury
Brief Title: SVF Combined With Functional Self-assembling Peptide Nanofiber Hydrogels in the Treatment of Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kunming Tongren Hospital (Industry)
Responsible Party: Principal Investigator, Hui Zhu, Director, Kunming Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KunmingTH_HZ_003
Record Dates: First submitted 2023-07-07; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Stromal Vascular Fraction (SVF) combined with Functional self-assembling peptide nanofiber hydrogels — Transplantation of SVF and biomimetic nanohydrogel

SUMMARY:
Traumatic spinal cord injury (SCI) is a severe medical problem experienced by people worldwide with high mortality and long term morbidity. Although progress has been made in understanding cellular and molecular mechanisms of SCI, treatment and management protocols aimed at ameliorating neurologic damage in patients remain ineffective. Cells and biomaterials offer new hope for the treatment of SCI.

Up to now, there have been many studies on the treatment of SCI using cells and biomaterials. Stromal Vascular Fraction (SVF) is a heterogeneous mixture of cells obtained from adipose tissue. These cells include adipose-derived stem cells, endothelial cells, endothelial progenitor cells, pericytes, T cells, and other immune cells. SVF has strong self-renewal, proliferation and differentiation potential, it can replace necrotic cells and synthesize a variety of bioactive factors through paracrine and autocrine, activate cell and vascular regeneration pathways. Therefore, SVF shows significant advantages. The sequence of functional self-assembling peptide nanofiber hydrogels (hereinafter referred to as hydrogels) is HGF(RADA)4RIKVAV (H: histidine; G: Glycine; F: phenylalanine; R: arginine; A: Alanine; D: aspartic acid; I: isoleucine; K: Lysine; V: valerine). The hydrogel is based on the short peptide RADA16 ((RADA)4, which is already available in the product PuramatrixTM for clinical hemostasis and cell culture, but the aqueous solution of PuramatrixTM is acidic which harms cells and tissues upon direct contact. While the hydrogels in this study is pH neutral and does not harm cells and tissues. Articles published by the provider demonstrate that hydrogels can support 3D stem cell growth, have good biocompatibility in vivo (animal spinal cord), and promote neural regeneration after SCI. The chemical structure of the hydrogels is simple and clear, and the degradation product is amino acid. Therefore, SVF and the hydrogel from functional self-assembling peptide are combined for SCI repair in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults, 18-60 years of age, with a clinical diagnosis of chronic traumatic SCI (≥ 3 months after SCI)
2. Neurological examination: ASIA-A
3. Both the spinal and neurological levels of injury were between T1-T12
4. Subjects must be able to read, write and complete visual analogue scale
5. Voluntarily signs and dates an informed Consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to any study-specific procedures.

Exclusion Criteria:

1. Subjects with osteoporosis or had joint disease
2. Severe head injury
3. Severe pressure sore
4. Sign of kidney, cardiovascular, liver disorders
5. Subjects with internal medical and/or infectious diseases (including but not limited to Hepatitis B and HIV carriers)
6. Pregnant women or women at lactation stages
7. Medically or mentally unstable according to the judgment of the investigator
8. History of multiple sclerosis or peripheral demyelination
9. Any criteria which, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Kunming Locomotor Scale (KLS) at 12 months | Day 0, Month 12
  Scale from minimum (1) to maximum (10), higher scales mean a better outcome.

SECONDARY OUTCOMES:
Change from Baseline Walking Index for Spinal Cord Injury at 12 months | Day 0, Month 12
  Score from minimum (0) to maximum (20), higher scores mean a better outcome.
Change from Baseline American Spinal Injury Association International Standards for Neurologic Classification of Spinal Cord Injury at 12 months | Day 0, Month 12
  Motor scores: bilateral upper and lower extremities total: minimum (0) to maximum (100), higher scores mean a better outcome.
  Sensory scores: bilateral light touch total from minimum (0) and maximum (112), bilateral pin prick from minimum (0) and maximum (112), higher scores mean a better outcome.
Change from Baseline Spinal Cord Independence Measure at 12 months | Day 0, Month 12
  Score from minimum (0) to maximum (100), higher scores mean a better outcome.
Change from Baseline Modified Ashworth Scale (MAS) at 12 months | Day 0, Month 12
  Scale from minimum (0) to maximum (4), higher scales mean a worse outcome.
Change from Baseline International Index of Erectile Function at 12 months | Day 0, Month 12
  Male subjects only. Score from minimum (0) to maximum (25), higher scores mean a better outcome.
Change from Baseline Numerical rating scale at 12 months | Day 0, Month 12
  Scale from minimum (0) to maximum (10), higher scales mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Kunming Tongren Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided